CLINICAL TRIAL: NCT04633746
Title: Validation of Plasma Endostatin for Predicting Renal Outcome From Acute Kidney Injury Induced by Sepsis
Brief Title: Plasma Endostatin Predicts Outcome of Septic AKI
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Farouk, clinical professor, Cairo University
Other Study IDs: I-801016
Record Dates: First submitted 2020-11-11; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Acute Kidney Injury Due to Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sepsis with AKI: Patients admitted with the diagnosis of sepsis associated with elevation of renal function tests
  Interventions: Diagnostic Test: measuring plasma Endostatin level
- Sepsis without AKI: Patients admitted with the diagnosis of sepsis with no elevation of renal function tests
  Interventions: Diagnostic Test: measuring plasma Endostatin level

INTERVENTIONS:
Diagnostic Test: measuring plasma Endostatin level — measuring plasma Endostatin level at the time of admission then after 48hrs and 96 hours

SUMMARY:
Introduction: Acute kidney injury (AKI) occurs up to 50% of patients admitted to intensive care unit. Plasma Endostatin, released from basement membrane of Bowman's capsule, rises early during AKI.

Aim of Work: To investigate the role of the plasma endostatin in the outcome prediction (renal recovery, ICU stay, mortality) of acute kidney injury in patients with sepsis.

Methods: a prospective, observational single center study on 40 patients with Sepsis at the Critical Care Department, Cairo University hospitals between March 2019 and November 2019. Serum plasma endostatin was measured at the day of admission & every 48hrs (3 samples). APACHE II, SOFA scores were calculated. Forced diuresis was used if indicated.

DETAILED DESCRIPTION:
The study was conducted on 40 patients with sepsis who admitted in the Critical Care department of Cairo University.

The sepsis is identified according to surviving sepsis campaign guidelines with use of SOFA score to establish the diagnosis.

The patients divided into 2 groups the first group included 25 patients who developed AKI as defined by KDIGO guidelines and the other group included 15 patients as a control group.

The Plasma Endostatin level is sampled in the first 24 hours of diagnosis of AKI, the estimation of plasma Endostatin level done by ELISA technique.

The results were presented in form of: descriptive, analytical and comparative data between the groups of study.

It was found that the patients with higher levels of plasma endostatin had a higher incidence of recovery from AKI and higher incidence of 28 days survival, while the patients with lower levels of plasma Endostatin below the determined Cut-off value have increased incidence of RRT .

Also that the patients with higher levels of plasma Endostatin levels were less labile to mechanical ventilation and had a higher incidence of weaning of vasopressors in comparison of the other group of lower levels of plasma Endostatin.

Plasma Endostatin levels have no difference between the AKI group and sepsis group which may need further investigations to determine its role in sepsis.

so that, the plasma Endostatin can be used as a marker of recovery from AKI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sepsis defined According to Surviving Sepsis Campaign 2016 sepsis: Suspected or documented infection in addition to increase in SOFA score 2 points or more from the baseline108.
* The patients will be followed for development of acute kidney injury (AKI) defined according to criteria established by Kidney Disease Improving Global Outcome guidelines (KDIGO) 20129 which includes any of the following criteria:

  * Increase in serum creatinine by > 0.3 mg/dl within 48 hours; or
  * Increase in serum creatinine to > 1.5 times baseline, which is Known or presumed to have occurred within the prior 7 days; or
  * Urine volume < 0.5 ml/kg/h for 6 hours.

Exclusion Criteria:

* Critically ill patients with known history of CKD.
* Patients on RRT ( intermittent or continuous)
* Post renal AKI.
* Not known history of nephrotoxic drug intake.
* Patient with contrast induced nephropathy
* Patients with cardiogenic shock who developed AKI.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age: 18- 80 years .
  - No gender preference
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Renal outcme | 7 days
  Number of participants who have recovered renal functions & those who needed Renal replacement therapy

CONTACTS AND LOCATIONS:
Overall Officials: farouk faris, Principal Investigator — Cairo University
Locations (1):
- Farouk Faris, Cairo, Down Town, Egypt

IPD SHARING:
Plan to Share IPD: No